CLINICAL TRIAL: NCT05074316
Title: A Prospective Registry Study on Biological Disease Profile, Intervention Type and Clinical Outcome in Patients With Myeloid Neoplasms
Brief Title: The Myeloid Neoplasms Biology and Outcome Project
Acronym: MyBOP
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard F Schlenk, Head of NCT trials center and Clinical Trials Office Hematology/Oncology, University Hospital Heidelberg
Other Study IDs: MyBOP
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Myeloid Neoplasm
Keywords: outcome project; registry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — clinically and molecularly annotated biospecimens are collected and stored within the biobank structures of the Department of Internal Medicine V of the Heidelberg University Hospital including blood and bone marrow samples, plasma and serum including liquid biopsies (cfDNA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Myeloid Neoplasms Biology and Outcome Project (MyBOP) aims to establish a registry study for patients with myeloid neoplasms. It integrates clinical data, biological samples, socio-demographic information, long-term follow-up and patient reported outcomes in a structured manner for scientific purposes.

The ultimate benefits are:

1. Improvement of evidence-based clinical management of patients with myeloid neoplasms through better understanding of the course of disease and prognostic and predictive parameters
2. Direct access to new and personalized treatment approaches through recruitment into clinical studies based on the myeloid neoplasms study platform
3. Quality assurance of participating centers by evaluating and comparing clinical outcomes and side effects of the MyBOP patients with published data.

DETAILED DESCRIPTION:
During recent years, considerable progress has been made in deciphering the molecular genetic and epigenetic basis of myeloid neoplasms and in defining new diagnostic and prognostic as well as predictive markers. Myeloid neoplasms are categorized according to the current WHO Classification of Tumors of Haematopoietic and Lymphoid Tissues based on the revision of 2016 [1]. This includes Myeloproliferative neoplasms (MPN), Mastocytosis, Myeloid/lymphoid neoplasms with eosinophilia and rearrangement of PDGFRA, PDGFRB, or FGFR1, or with PCM1-JAK2, Myelodysplastic/myeloproliferative neoplasms (MDS/MPN), Myelodysplastic syndromes (MDS), Myeloid neoplasms with germ line predisposition, Acute myeloid leukemia (AML) and related neoplasms (i.e. Myeloid sarcoma and Myeloid proliferations related to Down syndrome), Blastic plasmacytoid dendritic cell neoplasm and Acute leukemia of ambiguous lineage (Table 1).

A growing number of recurring genetic changes are recognized in the current WHO 2016 classification of myeloid neoplasms [2] and additional molecularly defined subgroups as well as new entities are expected to be included in future versions. Furthermore, novel therapies are now available and being developed, which target specific genetic lesions, and several surface antigens are being explored as targets for immunotherapy-based treatment strategies, e.g. CAR-T-cell therapy [3].

Although the WHO 2016 classification represents an enormous progress in terms of reliability, validity and objectivity, there are still huge diagnostic uncertainties left [4-18] and the field of targeted therapy [19-25] in myeloid neoplasms is just at its beginning. Furthermore, clonal evolution and transition from one entity to another is a clinically relevant issue [26-30].

Thus, key areas of interest are:

* Systematic collection and evaluation of comprehensive clinical information from patients with myeloid neoplasm, including morphomolecular disease subtype, as well as drug treatments, radiation therapy, surgical procedures and long-term follow-up data
* Systematic collection and evaluation of comprehensive biological specimens and information from patients with myeloid neoplasms, including data on the genomic, transcriptomic, epigenomic and proteomic "landscapes" as well as expression of surface antigens of myeloid disease subtypes, to identify novel prognostic and predictive parameters as well as entry points for targeted therapeutic interventions
* Regular assessment of patient reported outcomes

The above challenges are ideally met by a registry study with a sufficient population size in order to answer relevant questions in rare cancer entities. The aim is to set up a registry study that covers systematic and comprehensive clinical data acquisition. In addition, the banking of tumor and germline samples from patients with myeloid neoplasms is intended by all patients. This resource will spur patient-oriented investigations into relationships between clinical and biological parameters in myeloid neoplasms and lay the groundwork for novel, molecular mechanism- and immunotherapy-based treatment approaches in poorly understood and difficult-to-treat subsets.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or proven diagnosis of Myeloid Neoplasms according to the WHO Classification of Tumors of Haematopoietic and Lymphoid Tissues
* Age ≥18 years
* Ability to understand the nature and individual consequences of the registry
* Written informed consent
* Subjects who are physically or mentally capable of giving consent

Exclusion Criteria:

Severe neurological or psychiatric disorder interfering with the ability to give written informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: the patient cohort will be selected from the University Hospital Heidelberg.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
median overall survival (mOS) | 5 years
  Time period of survival from date of diagnosis of myeloid neoplasy
overall survival (mOS) | 10 years
  Time period of survival from date of diagnosis of myeloid neoplasy
event free survival (EFS) | 5 years
  Time period of event free survival from date of diagnosis of myeloid neoplasy
progression free survival (PFS) | 5 years
  Time period of progression survival from date of diagnosis of myeloid neoplasy

SECONDARY OUTCOMES:
Questionnaire for the health- related quality of life QLQ-C30 | 5 years
  Standardized Quality of Life Assessment, Higher values are better
Questionnaire for physical, cognitive and emotional aspects of cancer-related fatigue QLQ-FA12 | 5 years
  Standardized Quality of Fatigue, Higher values are worse
Questionnaire for anxiety and depression PHQ-4 | 5 years
  Standardized Quality of anxiety and depression, Higher values are worse
Functional Assessment of Cancer Therapy Fact-Cog | 5 years
  Standardized Quality of cognitive function, Higher values are better
The Pittsburgh Sleep Quality Index PSQI | 5 years
  Standardized Quality of sleep, Higher values are worse

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Schlenk, M.D., Principal Investigator — University Hospital Heidelberg, Department of Internal Medicine V, German Cancer Research Center
Locations (1):
- UHHeidelberg, Heidelberg, Baden-Wurttemberg, Germany